CLINICAL TRIAL: NCT00587561
Title: Efficacy of Social Cognition Training in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JMF0005; D4628W
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; social cognition; cognition; treatment; outcome
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Social Cognition Interaction Training (Experimental): Will receive 20-26 sessions of a manualized group treatment called Social Cognition Interaction Training
  Interventions: Behavioral: Social Cognition Interaction Training
- 2 Wait List Control (Other): Wait list control; 6 months of treatment as usual followed by Social Cognition Interaction Training group
  Interventions: Behavioral: WLC

INTERVENTIONS:
Behavioral: Social Cognition Interaction Training — manualized group therapy
  Arms: 1 Social Cognition Interaction Training
Behavioral: WLC — wait-list control for 6 months, followed by the experimental group therapy
  Arms: 2 Wait List Control

SUMMARY:
The term social cognition refers to how social information is processed. Individuals with schizophrenia and schizoaffective disorder have been shown to have significant deficits in social cognition. Moreover, it has been speculated that these deficits may in turn have a negative impact on their overall functioning. Behavioral interventions targeting social cognition are just beginning to emerge, and there is a need to evaluate their efficacy.

Objectives:

This is a small trial evaluating the efficacy of social cognition interaction training (SCIT) an experimental behavioral treatment for improving social cognition in schizophrenia.

Research Design and Methodology:

Approximately 48 participants with schizophrenia-spectrum disorders will be randomized into one of two conditions: 1) a 20 to 24 session manualized social cognition interaction training group (SCIT), or 2) wait-list control. Pre-and post-group therapy assessments of symptoms, social cognition, basic cognition, and community function will be conducted. Data obtained from this study will allow us to determine the efficacy of SCIT training in improving symptom, cognitive, and functional measures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder
* Age between 18 and 65
* minimum of 30 days since discharge from last hospitalization
* minimum of 30 days since last change in psychiatric medications
* no housing changes in the past 30 days

Exclusion Criteria:

* current diagnosis of alcohol or substance abuse/dependence
* history of brain trauma or neurological disease
* mental retardation or developmental disability
* auditory or visual impairment that would interfere with study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Fiszdon, Ph.D., Principal Investigator — VA Connecticut Heathcare System and Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

REFERENCES:
- [Result] Fiszdon JM, Dixon HD, Davidson CA, Roberts DL, Penn DL, Bell MD. Efficacy of social cognition and interaction training in outpatients with schizophrenia spectrum disorders: randomized controlled trial. Front Psychiatry. 2023 Aug 4;14:1217735. doi: 10.3389/fpsyt.2023.1217735. eCollection 2023. PMID 37599886

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Our initial plan had been to recruit and enroll 48 participants. 67 volunteers were assessed for eligibility. Of those, 9 did not meet inclusion criteria and 7 declined to participate after learning more about the study. Our initial plan had been to randomized 48 volunteers however due to concerns about potential drop-out, we recruited and randomized 51 participants.
Groups:
- Intervention: Social cognition interaction training (0 - 6 months), then crossed-over to treatment as usual.
- Waitlist Control: Treatment as usual (0 - 6 months), then crossed-over to social cognition interaction training.
Period: Overall Study
Arm/Group | Intervention | Waitlist Control
Started | 25 | 26
Completed | 19 | 22
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Intervention: 20-26 sessions of a manualized group treatment called social cognition interaction training (0 - 6 months), then crossed-over to treatment as usual.
- Waitlist Control: 6 months of treatment as usual followed by Social Cognition Interaction Training
- Total: Total of all reporting groups
Arm/Group | Intervention | Waitlist Control | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.56 (10.97) | 49.96 (9.15) | 47.80 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Social Cognitive Measures
Description: change score for Facial Emotion Identification Task (FEIT), FEIT scores range from 0-19 with higher scores indicating better performance, higher change scores indicate greater improvement
Time Frame: 6 months - baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Social Cognition Interaction Training: social cognition training
- Waitlist Control: wait list control
Arm/Group | Social Cognition Interaction Training | Waitlist Control
Number analyzed (Participants) | 19 | 22
score on a scale | 0.11 (2.00) | -1.68 (2.57)

2. Secondary Outcome: Basic Cognitive Measures
Description: change score on Matrics Consensus Cognitive Battery (MCCB) 6 domain composite average t-score, t-score mean = 50 and SD=10, higher change scores indicate greater improvement; please note outcome is not a t-score itself but a change in t-score
Time Frame: 6 months - baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Cognition Interaction Training | Waitlist Control
Number analyzed (Participants) | 18 | 22
score on a scale | 1.61 (7.42) | 0.81 (5.30)

ADVERSE EVENTS:
Groups:
- Intervention Group: Social Cognition Interaction Training: First period of Intervention Group, social cognition interaction training from 0 -6 months.
- Intervention Group: Treatment As Usual: Second period of Intervention Group, treatment as usual after 6 months.
- Waitlist Control Group, Treatment As Usual: First period of Waitlist Control Group, treatment as usual from 0 - 6 months.
- Waitlist Control Group, Social Cognition Interaction Training: Second period of Waitlist Control Group, social cognition interaction training after 6 months.
Arm/Group | Intervention Group: Social Cognition Interaction Training | Intervention Group: Treatment As Usual | Waitlist Control Group, Treatment As Usual | Waitlist Control Group, Social Cognition Interaction Training
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/25 | 1/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/26 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group: Social Cognition Interaction Training (N=25) | Intervention Group: Treatment As Usual (N=25) | Waitlist Control Group, Treatment As Usual (N=26) | Waitlist Control Group, Social Cognition Interaction Training (N=26)
hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — psychiatric symptom exacerbation and hospitalization
hospitalization for suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) — hospitalization for symptom exacerbation with suicidal ideation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes